CLINICAL TRIAL: NCT02655159
Title: Retrospective Observational Study of Nab-paclitaxel (Abraxane®) Treatment in Patients With Metastatic Breast Cancer in Routine Clinical Practice
Brief Title: Study of Nab-paclitaxel (Abraxane®) Treatment in Patients With Metastatic Breast Cancer in Routine Clinical Practice
Acronym: AMBER
Status: Terminated | Type: Observational
Why Stopped: Given the infeasibility to achieve the study population together with the loss of originality in the scientific rationale, it was considered to cancel the study
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-CMM-2015-01
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Metastatic breast cancer; nab-paclitaxel; Abraxane; Observational; Retrospective; AMBER
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abraxane® treatment in patients with metastatic breast cancer: Patients diagnosed with HER2-negative MBC who have started treatment with nab-paclitaxel monotherapy no further than the third line of chemotherapy for metastatic disease during the past 3 years (2012-2014) and who give their consent to data collection.

SUMMARY:
This is a national, multicenter, retrospective, observational post-authorization study (EPA-OD) study. The study will be conducted by reviewing the medical records of patients up to the start of the study. In each case, only data from before the start of the study will be obtained in order to ensure they are retrospective in nature, thus reflecting the regular use of nab-paclitaxel in clinical practice and avoiding interference with the physician's clinical practice.

To ensure the observational nature of this study, these data will be collected whenever they are available in the patient's medical record, and so no diagnostic or therapeutic intervention outside regular clinical practice will be used.

DETAILED DESCRIPTION:
This is a national, multicenter, retrospective, observational post-authorization study (EPA-OD) study. Investigators will include all consecutive adult patients diagnosed with HER2-negative MBC who have started treatment with nab-paclitaxel monotherapy no further than the third line of chemotherapy for metastatic disease during the past 3 years (2012-2014). These patients must meet all the inclusion criteria and none of the exclusion criteria established in this protocol.

The primary objective is to describe the effectiveness of nab-paclitaxel in terms of response in early lines of chemotherapy for metastatic breast cancer in routine clinical practice.

This study plans to collect data retrospectively, provided they are available in the patient's medical record and according to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age.
* Confirmed diagnosis of MBC (stage IV).
* Breast adenocarcinoma confirmed histologically.
* HER2-negative according to the American Society of Clinical Oncology (ASCO) and Anatomical Pathology (CAP) criteria for the detection of HER2 in breast cancer.
* Patients who have started treatment with nab-paclitaxel monotherapy no further than the third line of chemotherapy for metastatic disease in HER2-negative breast cancer during the period 2012-2014 (3 years) and who have received at least one cycle of treatment.
* Ability to give informed consent, preferably in writing or orally in front of a witness, before the start of data collection (if it is able to be given).

Exclusion Criteria:

* Patients with any medical or psychological disorder which in the investigator's opinion might compromise the ability of the patient to give their informed consent.
* Patients who have received treatment with nab-paclitaxel combined with other chemotherapy agents or anti-angiogenic drugs or tumor-targeting drugs with anti-tumor activity.
* Patients who have taken part in any clinical trial (interventional) during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with HER2-negative MBC who have started treatment with nab-paclitaxel monotherapy no further than third-line chemotherapy for metastatic disease between 2012 and 2014 will be enrolled consecutively. In addition, patients must meet the selection criteria established in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 8 months
  The number of patients who achieve a complete response (CR) or partial response (PR) based on RECIST v1.1 criteria during treatment with nab-paclitaxel until disease progression, the end of treatment or the start of the study, whichever comes first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 8 months
  The number of patients who achieve a complete response (CR) or partial response (PR) during the first 3 treatment cycles with nab-paclitaxel and the corresponding 95% CI will be calculated.
Disease control rate (DCR) | Up to approximately 8 months
  The percentage of patients with complete response (CR), partial response (PR), or stable disease (SD) for at least 16 weeks, and the corresponding 95% confidence intervals (CI) will be calculated.
Time to disease progression (TTP) | Up to approximately 8 months
  Is defined as the time from the start of treatment with nab-paclitaxel to disease progression or death due to progression. TTP will be estimated by using the Kaplan-Meier method. The median and confidence interval for the median at 95% reliability (95% CI) will be calculated. In patients who show no disease progression or who have not died, the date of censoring may be the day on which the patient's death is documented, the day of the last follow-up assessment or the day of the last tumor assessment in case the foregoing is not available.
Progression-free survival (PFS) | Up to approximately 8 months
  Is defined as the time from the start of treatment with nab-paclitaxel to disease progression or death from any cause. PFS will be estimated by using the Kaplan-Meier method. Patients who have shown no disease progression or who have not died at the time of data collection will be censored on the date on which it was last known that no disease progression occurred. The date of censoring may be the day of the last follow-up assessment or the day of the last tumor assessment in case the foregoing is not available.
Overall survival (OS) | Up to approximately 8 months
  Is defined as the time from the start of treatment with nab-paclitaxel to death from any cause. OS will be estimated by using the Kaplan-Meier method. Patients who have not died at the time of data collection will be censored on the date on which they are last known to be alive. The date of censoring may be the day of the last follow-up assessment or the day of the last tumor assessment in case the foregoing is not available.
Adverse Events (AEs) | Up to approximately 8 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Pellín, MD, Study Director — Celgene Spain
Locations (19):
- Spain (19):
  - Complejo Hospitalario Jaén, Jaén, Andalusia
  - Hospital Clínico Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Burgos, Burgos, Castille and León
  - Hospital Clínico Salamanca, Salamanca, Castille and León
  - Hospital Clínico Valladolid, Valladolid, Castille and León
  - Hospital Virgen Salud, Toledo, Castille-La Mancha
  - Hospital Vall d´Hebron, Barcelona, Catalonia
  - Hospital Universitario San Joan Reus, Reus, Catalonia
  - Hospital Infanta Cristina, Badajoz, Extremadura
  - Capio Clideba, Badajoz, Extremadura
  - Complejo Hospitalario Orense, Ourense, Galicia
  - Hospital Gregorio Marañón, Madrid, Madrid
  - MD Anderson, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 octubre, Madrid, Madrid
  - Hospital Quirón, Madrid, Madrid
  - Hospital Santa Lucía, Cartagena, Murcia
  - Hospital Morales Meseguer, Murcia, Murcia
  - Hospital Navarra, Pamplona, Navarre